CLINICAL TRIAL: NCT01221402
Title: Effect of Extended-Release Niacin on Saphenous Vein Graft Atherosclerosis: The Atherosclerosis Lesion Progression Intervention Using Niacin Extended Release in Saphenous Vein Grafts (ALPINE-SVG) Pilot Trial
Brief Title: Effect of Extended-Release Niacin on Saphenous Vein Graft Atherosclerosis
Acronym: ALPINE-SVG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-029; R01HL102442 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Aortocoronary Saphenous Vein Bypass Graft Atherosclerosis; Intermediate Saphenous Vein Graft Lesions
MeSH Terms: interventions — Niacin

STUDY DESIGN:
Intervention Model Description: Original plan was to enroll 138 subjects, but trial was terminated early and total randomized was 38.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-release niacin (Experimental)
  Interventions: Drug: extended-release niacin (Niaspan)
- Placebo (Placebo Comparator)
  Interventions: Drug: extended-release niacin (Niaspan)

INTERVENTIONS:
Drug: extended-release niacin (Niaspan) — Patients will be randomized in a 1:1 ratio to receive extended-release niacin (1500 - 2000 mg per day) or matching placebo that contains 50 mg of crystalline niacin (enough to cause flushing but has no effect on lipid levels).

SUMMARY:
Intermediate saphenous vein graft (SVG) lesions are common, have high rates of progression to severe lesions or occlusion, and are associated with high incidence of adverse clinical outcomes.

The ALPINE-SVG trial is a randomized-controlled trial of extended-release niacin vs. placebo in patients with intermediate saphenous vein graft lesions. The main hypothesis of the study is that compared to placebo, niacin administration will result in reduction in percent atheroma volume at 12-month follow-up angiography.

DETAILED DESCRIPTION:
This is a phase II, single-center, double-blind trial that will randomize 138 prior CABG patients with an intermediate SVG lesion (30%-60% angiographic diameter stenosis) on clinically-indicated coronary angiography, and HDL-C<60 mg/dL to ER-niacin at a dose of 1500-2000 mg daily or matching placebo (containing 50 mg of niacin that can cause flushing but has no lipid lowering effect) for 12 months. All patients will receive a statin with goal LDL-C <70 mg/dL. Coronary angiography, intravascular ultrasonography (IVUS), and intravascular near-infrared intracoronary spectroscopy (NIRS), and optical coherence tomography (OCT) of the intermediate SVG lesion will be performed at enrollment and after 12 months in each patient, along with exercise stress testing at 1 month and 12 months, B-mode carotid ultrasound imaging at enrollment and after 6 and 12 months, reactive hyperemia peripheral arterial tonometry (RH-PAT) at enrollment and after 6 and 12 months, and with peripheral blood sampling performed at enrollment and at 1, 3, 6, 9 and 12 months, to determine whether compared to placebo, administration of ER-niacin will result in:

1. Reduction of the percent atheroma volume (PAV) of the intermediate SVG lesion at 12-month follow-up IVUS imaging (primary endpoint)
2. Reduction of total and normalized total intermediate SVG lesion atheroma volume, reduction of atheroma volume in the most diseased 10-mm subsegment of the target intermediate lesion, reduction of atheroma volume in the subsegment of the target intermediate lesion with lipid core plaque by NIRS, reduction of lipid core burden index as assessed by near-infrared intracoronary spectroscopy, increase in fibrous cap thickness and reduction in the prevalence and number of microchannels, in the presence and extent of necrotic lipid pool, plaque rupture, calcification, and thrombus, as assessed by optical coherence tomography, and reduction of angiographic intermediate SVG target lesion failure at 12-month follow-up SVG imaging (secondary endpoints)
3. Increased exercise capacity and reduction in ischemia, as assessed by exercise stress testing between 1 and 12 months (secondary endpoint)
4. Less increase in mean carotid intima-media thickness at 6 and 12 months (secondary endpoint)
5. Greater increase in natural logarithmic scaled reactive hyperemia index (L_RHI) at 6 and 12 months (secondary endpoint)
6. Greater increase in EPC-CFU/mL of peripheral blood from baseline to 1, 3, 6, and 12 months post enrollment (secondary endpoint)
7. Reduction of major adverse cardiac events (defined as the composite of death, acute coronary syndrome, or coronary revascularization) during follow-up (secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater
2. Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
3. Undergoing clinically-indicated coronary and SVG angiography
4. Have an intermediate SVG lesion (defined as a lesion 30-60% angiographic diameter stenosis) without previous percutaneous intervention, amenable to examination with IVUS. The lesion should have no thrombus or ulceration and should not be considered responsible for the patient's clinical presentation and referral for graft angiography.

Exclusion Criteria:

1. Known allergy to niacin
2. History of statin-induced myopathy
3. Positive pregnancy test or breast-feeding
4. Coexisting conditions that limit life expectancy to less than 12 months or that could affect a patient's compliance with the protocol
5. Uncontrolled fasting triglyceride levels ( 500 mg/dL)
6. Fasting LDL-C >200 mg/dL
7. Fasting HDL-C >60 mg/dL
8. Poorly controlled diabetes (glycosylated hemoglobin levels 10%)
9. Current active liver disease or hepatic dysfunction
10. AST or ALT > 2x the upper limit of normal
11. Uncontrolled hypothyroidism (Thyroid Stimulating Hormone >1.5 x upper limit of normal [ULN])
12. Unexplained creatine kinase elevations (>3 x ULN)
13. Recent history of acute gout
14. Serum creatinine > 2.5 mg/dL
15. HIV (due to potential anti-retroviral drug-interactions with niacin)
16. Use of high-dose, antioxidant vitamins (vitamins C, E, or beta-carotene) that may interfere with the HDL-raising effect of niacin
17. Severe peripheral arterial disease limiting vascular access
18. Referral for cardiac catheterization by a physician who is an investigator in the present study.
19. Symptoms consistent with moderate or greater severity of congestive heart failure (New York Heart Association - NYHA class III or IV) or whose most recent determination of left ventricular ejection fraction is <25%
20. Uncontrolled hypertension, defined as either a resting diastolic blood pressure of ≥100 mmHg or a resting systolic blood pressure of ≥200 mmHg
21. History of allergic reaction to iodine-based contrast agents
22. Significant medical or psychological condition that, in the opinion of the investigator, may compromise the patient's safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
change in percent atheroma volume at 12 months intravascular ultrasonography | 12 months

SECONDARY OUTCOMES:
change in total and normalized total intermediate SVG lesion atheroma volume | 12 months
reduction of atheroma volume in the most diseased 10-mm subsegment of the target intermediate lesion | 12 months
reduction of atheroma volume in the subsegment of the target intermediate lesion with lipid core plaque by near-infrared spectroscopy | 12 months
lipid core burden index as assessed by near-infrared intracoronary spectroscopy | 12 months
increase in fibrous cap thickness and reduction in the prevalence and number of microchannels, in the presence and extent of necrotic lipid pool, plaque rupture, calcification, and thrombus, as assessed by optical coherence tomography | 12 months
angiographic intermediate SVG target lesion failure | 12 month
exercise capacity and ischemia, as assessed by exercise stress testing | 12 months
carotid intima-media thickness | 6 and 12 months
reactive hyperemia index | 12 months
EPC-CFU/mL of peripheral blood | 12 months
major adverse cardiac events (defined as the composite of death, acute coronary syndrome, or coronary revascularization) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Healthcare System, Dallas, Texas, United States

REFERENCES:
- [Result] Kotsia AP, Rangan BV, Christopoulos G, Coleman A, Roesle M, Cipher D, de Lemos JA, McGuire DK, Packer M, Banerjee S, Brilakis ES. Effect of Extended-Release Niacin on Saphenous Vein Graft Atherosclerosis: Insights from the Atherosclerosis Lesion Progression Intervention Using Niacin Extended Release in Saphenous Vein Grafts (ALPINE-SVG) Pilot Trial. J Invasive Cardiol. 2015 Oct;27(10):E204-10. PMID 26429851
- [Result] Guerra A, Rangan BV, Coleman A, Xu H, Kotsia A, Christopoulos G, Sosa A, Chao H, Han H, Abdurrahim G, Roesle M, de Lemos JA, McGuire DK, Packer M, Banerjee S, Brilakis ES. Effect of Extended-Release Niacin on Carotid Intima Media Thickness, Reactive Hyperemia, and Endothelial Progenitor Cell Mobilization: Insights From the Atherosclerosis Lesion Progression Intervention Using Niacin Extended Release in Saphenous Vein Grafts (ALPINE-SVG) Pilot Trial. J Invasive Cardiol. 2015 Dec;27(12):555-60. PMID 26630643